CLINICAL TRIAL: NCT04958746
Title: A Multi-Center, Randomized, Double-Blind, Propofol Parallel-Controlled Phase III Clinical Trial Evaluating the Efficacy and Safety of Ciprofol Injection for the Induction of Sedation/Anesthesia in Subjects Undergoing Gynecological Outpatient Surgeries
Brief Title: Phase III Clinical Trial Evaluating the Efficacy and Safety of Ciprofol Injection for the Induction of Sedation/Anesthesia in Subjects Undergoing Gynecological Outpatient Surgeries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK3486-308
Record Dates: First submitted 2021-06-23; First posted 2021-07-12 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Gynecological Outpatient Surgery
MeSH Terms: interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciprofol (Experimental): Ciprofol group：0.4/0.2mg/kg
  Interventions: Drug: Ciprofol
- Propofol (Placebo Comparator): Propofol group：2.0/1.0mg/kg
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Ciprofol — intravenous bolus
  Arms: Ciprofol
Drug: Propofol — intravenous bolus
  Arms: Propofol

SUMMARY:
This study is a multi-center, randomized, double-blind, Propofol parallel-controlled phase III clinical study, with the primary objective of evaluating the efficacy of Ciprofol vs. Propofol for the induction of sedation/anesthesia in subjects undergoing gynecological outpatient surgeries and secondary objective of evaluating the safety of Ciprofol in subjects undergoing gynecological outpatient surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. Patient needing gynecological outpatient surgery under general anesthesia without endotracheal intubation;
2. Female, aged between 18-65 (inclusive);
3. American Society of Anesthesiologists (ASA) Class I- II
4. Body mass index (BMI) ≥ 18 and ≤ 30 kg/m2;
5. Vital signs during the screening period meet the following criteria:

   1. Respiratory rate ≥ 10 and ≤ 24 breaths/min;
   2. Pulse oxygen saturation (SpO2) ≥ 95% when inhaling;
   3. Systolic blood pressure (SBP) ≥ 85 mmHg and ≤ 140 mmHg;
   4. Diastolic blood pressure (DBP) ≥ 50 mmHg and ≤ 90 mmHg;
   5. Heart rate ≥ 50 beats/min and ≤ 100 beats/min. (Note: For heart rate, the heart rate results of 12-ECG examination are used as the basis for judging whether the inclusion criteria are met.)
6. Capable of understanding the procedure and method of this study, willing to sign an informed consent form and to complete this study in strict accordance with the study protocol.

Exclusion Criteria:

1. Patients with contraindications to deep sedation/general anesthesia or a history of past sedation/anesthesia accidents;
2. Known sensitivity to Propofol Injection, Ciprofol Injection, the excipients in the investigational drugs (soybean oil, glycerin, triglyceride, egg lecithin, purified lecithin, sodium oleate, sodium hydroxide and disodium edetate), and opioids or any ingredient of opioids; contraindications to Propofol;
3. Patients with positive urine HCG or blood HCG (except abortion, dilatation and curettage, other outpatient surgeries for termination of pregnancy);
4. Patients having the following medical history or evidence prior to screening, which may increase sedation/anesthesia risk:

   1. History of cardiovascular diseases: Uncontrolled hypertension or SBP > 140 mmHg and/or DBP > 90 mmHg despite antihypertensive treatment, severe arrhythmia, heart failure, Adams-Stokes syndrome, unstable angina, myocardial infarction within 6 months prior to screening, history of tachycardia/bradycardia requiring medication, third-degree atrioventricular block or QTcF interval ≥ 450 ms (Fridericia's correction formula) during screening;
   2. Respiratory system disorders: Respiratory insufficiency, history of obstructive pulmonary disease, history of bronchospasm requiring treatment within 3 months prior to screening, acute respiratory tract infection with any one of the obvious symptoms such as fever, wheezing, or productive cough within 1 week prior to screening;
   3. History of neurological and mental disorders: history of craniocerebral injury, convulsions, epilepsy, intracranial hypertension, cerebral aneurysm, or cerebrovascular accident; history of schizophrenia, mania, chronic use of antipsychotics, cognitive impairment, etc.;
   4. History of gastrointestinal diseases: history of gastrointestinal retention, active hemorrhage, gastroesophageal reflux or obstruction, etc. which may cause reflux and aspiration, as per the judgment of the investigator;
   5. History of uncontrolled and clinically significant diseases in such as liver, kidney, blood system, nervous system, or metabolic system judged by the investigator to be unsuitable for this trial;
   6. History of alcohol abuse within 3 months prior to screening, abuse defined as average of > 2 units of alcohol per day (1 unit = 360 mL of beer or 45 mL of liquor with 40% alcohol or 150 mL of wine);
   7. History of drug abuse within 3 months prior to screening;
   8. Serious infection, trauma, or major surgery within 4 weeks prior to screening.
5. Patients with the following airway management risks at screening:

   1. Asthma history, and stridor;
   2. Sleep apnea syndrome;
   3. History or family history of malignant hyperthermia;
   4. History of intubation failure;
   5. Judged by the investigator to have difficult airway or judged as difficult tracheal intubation (modified Mallampati score III or IV).
6. Receiving any one of the following medications or treatments at screening:

   1. Participated in other clinical trials of drugs within 1 month prior to screening;
   2. Used Propofol, other general sedatives/anesthetics, and/or opioid analgesics or compounds containing opioid analgesics within 3 days prior to screening.
7. Patient whose laboratory parameters measured at screening meet any of the following criteria and are verified through reexamination:

   1. Neutrophil count < 1.5 × 109/L;
   2. Platelet count < 80 × 109/L;
   3. Hemoglobin < 90 g/L;
   4. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3.0 × upper limit of normal (ULN)
   5. Total bilirubin > 2 × ULN;
   6. Serum creatinine > 1.5 × ULN.
8. Breastfeeding females; women of child-bearing potential who are unwilling to use contraception during the trial; or subjects who are planning pregnancy within 1 month after completion of the trial.
9. Subject judged by the investigator to have any other factors unsuitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Success rate of anesthesia | Day 1
  The proportion of subjects successfully anesthetized in all subjects of the group.

SECONDARY OUTCOMES:
Time to successful sedation/anesthetic induction | Day 1
  Time from the initial administration of the investigational drug to the first time when MOAA/S is ≤ 1
Time to full recovery: | Day 1
  Time from the last administration of the investigational drug to the first of 3 consecutive MOAA/S scores = 5
Time to discharge | Day 1
  The time from the last administration of the investigational products to the first of 3 consecutive Aldrete scores of ≥ 9
Sedation/anesthesia satisfaction, including satisfaction evaluation of subjects, anesthesiologists, and surgeons. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Dongxin Wang, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China

REFERENCES:
- [Derived] Xu J, Yang M, Zeng Y, Zou XH, Ren JH, Xia Z, Xie HH, Yu YH, Xu MJ, Chen W, Wang DX. Efficacy and safety of ciprofol for sedation in outpatient gynecological procedures: a phase III multicenter randomized trial. Front Med (Lausanne). 2024 Apr 23;11:1360508. doi: 10.3389/fmed.2024.1360508. eCollection 2024. PMID 38716419